CLINICAL TRIAL: NCT05971797
Title: Rational-emotional Behavioral Therapy in Patients With Osteoarthritis and Concomitant Diseases Before Knee or Hip Arthroplasty
Brief Title: Rational-emotional Behavioral Therapy (REBT) in Patients With Osteoarthritis and Concomitant Diseases Before Arthroplasty
Acronym: REBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Organization, Federal Center for Traumatology, Orthopedics and Arthroplasty (Other)
Collaborators: Chuvash State University named after I.N. Ulyanov (Unknown)
Responsible Party: Principal Investigator, Emelianov Vladimir, MD PhD Clinical Assistant Professor, Federal State Budgetary Organization, Federal Center for Traumatology, Orthopedics and Arthroplasty
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2020-9
Record Dates: First submitted 2023-07-05; First posted 2023-08-02 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Depression, Anxiety; Pain
Keywords: Depression; Anxiety; Rational Emotive Behavior Therapy; Arthroplasty; Osteoarthritis; Comorbidities
MeSH Terms: conditions — Depression; Anxiety Disorders; Pain; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial in patients with depression or anxiety identified at prior psychological counseling prior to joint replacement surgery with or without comorbidities
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Comorbidities (Experimental): Upon admission to the hospital for surgery to replace large joints (knee or hip joints) and diagnosis with osteoarthritis of the knee or hip joint (M15.0, M16, M17), patients with comorbidities underwent 20-minute psychological counseling (PC) session. During PC the levels of depression (F32.0, F32.1 or F32.9) and anxiety (F41.0, F41.1, F41.3, F41.8 or F41.9) were assessed using the STAI and HADS questionnaires. In the experimental group, patients with identified increased levels of depression or anxiety underwent a session of rational-emotional-behavioral therapy, which aimed to modify incorrect thinking patterns. The level of anxiety and depression was reassessed after the surgery.
  Interventions: Behavioral: REBT
- Comorbidities control (No Intervention): Upon admission to the hospital for surgery to replace large joints (knee or hip joints) and diagnosis with osteoarthritis of the knee or hip joint (M15.0, M16, M17), patients with comorbidities underwent 20-minute PC. During PC, their levels of depression (F32.0, F32.1 or F32.9) and anxiety (F41.0, F41.1, F41.3, F41.8 or F41.9) were assessed using the STAI and HADS questionnaires. In the first control group, patients with identified increased levels of depression or anxiety did not receive REBT therapy. The level of anxiety and depression was reassessed after the surgery.
- No comorbidities (Active Comparator): Upon admission to the hospital for surgery to replace large joints (knee or hip joints) and diagnosis with osteoarthritis of the knee or hip joint (M15.0, M16, M17), patients without comorbidities underwent 20-minute PC session. During PC the levels of depression (F32.0, F32.1 or F32.9) and anxiety (F41.0, F41.1, F41.3, F41.8 or F41.9) were assessed using the the STAI and HADS questionnaires. In the second control group, patients with identified increased levels of depression or anxiety underwent a session of rational-emotional-behavioral therapy, which aimed to modify incorrect thinking patterns. The level of anxiety and depression was reassessed after the surgery.
  Interventions: Behavioral: REBT

INTERVENTIONS:
Behavioral: REBT — During REBT in patients with osteoarthritis and concomitant diseases with diagnosed depression or anxiety before arthroplasty the patients learn how to manage their irrational or unhealthy emotions, thoughts, and behaviors.
  Arms: Comorbidities; No comorbidities

SUMMARY:
The objective of this study was evaluation of the effectiveness of REBT on the emotional state of orthopedic patients with comorbidities before and after arthroplasty.

DETAILED DESCRIPTION:
The studies assessed depression or anxiety in orthopedic patients by using Spielberger State-Trait Anxiety Inventory (STAI) and Hospital Anxiety and Depression Scale (HADS) before and after athroplasty. The comorbid background studied. The orthopedic patients with comorbidities were divided into several groups: arterial hypertension, chronic pyelonephritis , varicose veins, cardiovascular disease and atherosclerosis, diabetes mellitus, infection diseases, gastrointestinal diseases, obesity, neurological disorder, cerebrovascular accident, iron deficiency anemia, chronic bronchitis, hyperthyroidism, cardiac arrhythmia, other diseases. Patients with high levels of anxiety and depression underwent Rational Emotive Behavior Therapy before surgery. Patients without comorbidities and patients with comorbidities but without exposure considered as a control.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled for the primary knee or hip arthroplasty (M15.0, M16, M17) before operation.

Exclusion Criteria:

* Other types of psychiatric pathology
* Reluctance to undergo psychological correction
* Failure to pass pre-test
* Ongoing follow-up with a psychologist or psychiatrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
STAI | 2 days after surgery
  Each subscale uses a 4-point Likert scale with a range from 1 ("not at all" for S- or "almost never" for T-Anxiety) to 4 ("very much so" for S- and "almost always" for T-Anxiety). Reverse scoring is used for anxiety-absent items (e.g., "I feel calm" or "I am happy"), and therefore, a higher score indicates more severe anxiety with a potential range from 20 to 80 for each subscale. According to the developer scores of 20-39, 40-59, and 60-80 indicate low, moderate, and high anxiety, respectively. Normative values are available in the manual.
HADS | 2 days after surgery
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). with a range from 0 ("not at all") to 3 ("most of the time"). Reverse scoring is used for items with positive wording (e.g., "I still enjoy the things I used to enjoy"). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). A score of 8-10 should be classified as a mild disorder, 11-15 as a moderate disorder, and 16 or more as a severe disorder.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Center for Traumatology, Orthopedics and Endoprosthetics, Cheboksary, Chuvashskaya Respublika, Russia